CLINICAL TRIAL: NCT05124457
Title: A Phase 2 Open Label Randomized Controlled Trial Determir Vs Neutral Protamine Hagedorn (NPH) In Pregnant Women: DETERMINE Study
Brief Title: DETERMINE: Detemir vs NPH
Acronym: DETERMINE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Christina S. Han, Maternal-Fetal Medicine Division Director, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DETERMINE
Record Dates: First submitted 2021-10-25; First posted 2021-11-18 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Gestational Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Intervention Model Description: Randomization to receive either insulin NPH or insulin detemir
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin Detemir (Experimental): Patients are to receive insulin detemir as long acting insulin to control blood sugars
  Interventions: Drug: Insulin Detemir
- Insulin NPH (Active Comparator): Patients are to receive insulin NPH as long acting insulin to control blood sugars
  Interventions: Drug: Insulin NPH

INTERVENTIONS:
Drug: Insulin Detemir — Patients are to receive insulin detemir
  Arms: Insulin Detemir
Drug: Insulin NPH — Patients are to receive insulin NPH
  Arms: Insulin NPH

SUMMARY:
The purpose of the study is to compare rates of neonatal hypoglycemia with maternal NPH vs determir use.

DETAILED DESCRIPTION:
Insulin detemir has been used and is FDA approved for type 1 diabetes in pregnancy women and its safety has been well established. At this point, the only long or intermediate acting medication that is approved for type 2 diabetes or gestational diabetes is insulin NPH. The most serious side effect of insulin detemir is hypoglycemia but the rates of hypoglycemia are lower when comparted to NPH both during pregnancy and outside of pregnancy. Diabetes mellitus (DM) is the most common diagnosis in pregnancy and its incidence is continuing to increase. Recent epidemiologic reports place the risk of pre-gestational diabetes at 1-2% and gestational diabetes (GDM) at 12.5%. Risk factors for type 2 diabetes (T2DM) and GDM include obesity, hypertension, family history of diabetes, polycystic ovarian syndrome, or excessive weight gain in pregnancy. Suboptimal control of DM in pregnancy confers significant morbidity on both the mother and fetus, including increased risk of preeclampsia, preterm delivery, perineal lacerations, cesarean delivery, neonatal hypoglycemia, and NICU admissions.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include pregnant women with pre-existing T2DM and GDM who requiring insulin to manage their blood sugars in pregnancy.

Exclusion Criteria:

1. Multiple Gestation
2. Type 1 Diabetes mellatus
3. Age < 18
4. Known or suspected hypersensitivity to NPH or insulin detemir
5. Known fetal major malformations
6. Chronic renal or hepatic insufficiency
7. Known to be HIV, Hepatitis B, or Hepatitis C positive
8. Indication for planned premature delivery (placenta accrete, or prior classical cesarean delivery)
9. Insulin dependent before conception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Neonatal Hypoglycemia | Within the first 24 hours of life
  Rate (%) of neonatal hypoglycemia
Prolonged neonatal hypoglycemia | Neonatal hypoglycemia after the 1st 24 hours of life but before discharge
  Rate (%) of prolonged neonatal hypoglycemia

SECONDARY OUTCOMES:
Neonatal Gastrin Level | At birth
  Sample form cord blood
Neonatal C-Peptide Level | At birth
  Sample from cord blood
Neonatal insulin level | At birth
  Sample from cord blood
Neonatal leptin level | At birth
  Sample from cord blood
Rates of pregnancy induced hypertension | 1 year
  Maternal rates of preeclampsia, eclampsia, or gestational hypertension
Mode of delivery | At delivery
  Spontaneous vaginal, operative vaginal, cesarean
Gestational Age at delivery | At delivery
  Gestational Age at delivery
Maternal glycemic control | 1 year
  Rate (%) of in range maternal blood glucose control in antepartum period
Total daily insulin | 1 year
  Total daily insulin dose in patient
Fetal anomolies | At birth
  Rate (%) of fetal anomolies
Macrosomia | At birth
  Rate (%) of macrosomia
Polyhydramnios | At birth
  Rate (%) of polyhydramnios
Neonatal weight | At birth
  Neonatal weight
Need for supplemental oxygen | 1 year
  Rate of supplemental oxygen use (%) in neonate
Need for dextrose infusion in neonate | 1 year
  Rate of dextrose infusion use (%) in neonate
Rates of respiratory distress syndrome | 1 year
  Rate of RDS (%) in neonate
5 Minute APGAR | At birth
  5 Minute APGAR

CONTACTS AND LOCATIONS:
Overall Officials: Christina Han, MD, Principal Investigator — University of California, Los Angeles; Michael Richley, MD, Study Director — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coton SJ, Nazareth I, Petersen I. A cohort study of trends in the prevalence of pregestational diabetes in pregnancy recorded in UK general practice between 1995 and 2012. BMJ Open. 2016 Jan 25;6(1):e009494. doi: 10.1136/bmjopen-2015-009494. PMID 26810997
- [Background] Melchior H, Kurch-Bek D, Mund M. The Prevalence of Gestational Diabetes. Dtsch Arztebl Int. 2017 Jul 16;114(24):412-418. doi: 10.3238/arztebl.2017.0412. PMID 28669379
- [Background] Mathiesen ER, Hod M, Ivanisevic M, Duran Garcia S, Brondsted L, Jovanovic L, Damm P, McCance DR; Detemir in Pregnancy Study Group. Maternal efficacy and safety outcomes in a randomized, controlled trial comparing insulin detemir with NPH insulin in 310 pregnant women with type 1 diabetes. Diabetes Care. 2012 Oct;35(10):2012-7. doi: 10.2337/dc11-2264. Epub 2012 Jul 30. PMID 22851598
- [Background] Hirsch IB, Juneja R, Beals JM, Antalis CJ, Wright EE. The Evolution of Insulin and How it Informs Therapy and Treatment Choices. Endocr Rev. 2020 Oct 1;41(5):733-55. doi: 10.1210/endrev/bnaa015. PMID 32396624
- [Background] Herrera KM, Rosenn BM, Foroutan J, Bimson BE, Al Ibraheemi Z, Moshier EL, Brustman LE. Randomized controlled trial of insulin detemir versus NPH for the treatment of pregnant women with diabetes. Am J Obstet Gynecol. 2015 Sep;213(3):426.e1-7. doi: 10.1016/j.ajog.2015.06.010. Epub 2015 Jun 9. PMID 26070699
- [Background] Dalgic N, Ergenekon E, Soysal S, Koc E, Atalay Y, Gucuyener K. Transient neonatal hypoglycemia--long-term effects on neurodevelopmental outcome. J Pediatr Endocrinol Metab. 2002 Mar;15(3):319-24. doi: 10.1515/jpem.2002.15.3.319. PMID 11924935
- [Background] O'Neill SM, Kenny LC, Khashan AS, West HM, Smyth RM, Kearney PM. Different insulin types and regimens for pregnant women with pre-existing diabetes. Cochrane Database Syst Rev. 2017 Feb 3;2(2):CD011880. doi: 10.1002/14651858.CD011880.pub2. PMID 28156005
- [Background] Kadakia R, Talbot O, Kuang A, Bain JR, Muehlbauer MJ, Stevens RD, Ilkayeva OR, Lowe LP, Metzger BE, Newgard CB, Scholtens DM, Lowe WL; HAPO Study Cooperative Research Group. Cord Blood Metabolomics: Association With Newborn Anthropometrics and C-Peptide Across Ancestries. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4459-4472. doi: 10.1210/jc.2019-00238. PMID 31498869
- [Background] Lowe WL Jr, Bain JR, Nodzenski M, Reisetter AC, Muehlbauer MJ, Stevens RD, Ilkayeva OR, Lowe LP, Metzger BE, Newgard CB, Scholtens DM; HAPO Study Cooperative Research Group. Maternal BMI and Glycemia Impact the Fetal Metabolome. Diabetes Care. 2017 Jul;40(7):902-910. doi: 10.2337/dc16-2452. PMID 28637888
- [Background] Fishel Bartal M, Ward C, Blackwell SC, Ashby Cornthwaite JA, Zhang C, Refuerzo JS, Pedroza C, Lee KH, Chauhan SP, Sibai BM. Detemir vs neutral protamine Hagedorn insulin for diabetes mellitus in pregnancy: a comparative effectiveness, randomized controlled trial. Am J Obstet Gynecol. 2021 Jul;225(1):87.e1-87.e10. doi: 10.1016/j.ajog.2021.04.223. Epub 2021 Apr 15. PMID 33865836
- [Background] Chun J, Strong J, Urquhart S. Insulin Initiation and Titration in Patients With Type 2 Diabetes. Diabetes Spectr. 2019 May;32(2):104-111. doi: 10.2337/ds18-0005. PMID 31168280
- See also: Abstract — https://doi.org/10.1016/j.ajog.2019.11.450
- See also: Abstract — https://doi.org/10.1016/j.ajog.2019.11.057